CLINICAL TRIAL: NCT07353918
Title: Neuromodulation Using Low-intensity Focused Ultrasound for Potential Treatment for Medically Refractory Temporal Lobe Epilepsy
Brief Title: Low-Intensity Focused Ultrasound Neuromodulation for Epilepsy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Carilion Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-24-2194
Record Dates: First submitted 2025-12-22; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Epilepsy (Treatment Refractory); Epilepsy Comorbidities
Keywords: LIFU; Neuromodulation; Seizure
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Intervention Model Description: This study is a within subject cross-over design with 1 visit with a real LIFU application, and 1 visit with a sham LIFU application. Order will be randomized.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not know which visit is real and which is sham. Both appear identical to the participant. The sham is performed by blocking the energy applied to the skull during LIFU. Analysis will be done prior to unblinding researchers. Only researchers interacting with the participant will know visit order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- LIFU- real (Experimental): Low-intensity focused ultrasound will be applied to the entorhinal cortex in a pre/post design.
  Interventions: Device: Low-intensity Focused Ultrasound
- LIFU - Sham (Sham Comparator): Sham Low-intensity focused ultrasound will be applied to the entorhinal cortex in a pre/post design.
  Interventions: Device: Sham

INTERVENTIONS:
Device: Low-intensity Focused Ultrasound — focused ultrasound transducer.
  Arms: LIFU- real
Device: Sham — Sham application of LIFU - energy blocked. Targeted to the same target as intervention.
  Arms: LIFU - Sham

SUMMARY:
This study is an invite only study looking at the effects of Low-Intensity Focused Ultrasound (LIFU) on epilepsy patients with implanted electrodes under the care of Dr. Shah.

DETAILED DESCRIPTION:
This project will explore the use of Low-Intensity Focused Ultrasound (LIFU) as a non-invasive method to reduce seizures and potentially enhance cognitive functions in epilepsy patients. LIFU can target specific deep brain areas without surgery, offering an alternative to invasive procedures. The study focuses on patients who have an implanted Responsive Neurostimulation System (RNS). LIFU will be used to stimulate the entorhinal cortex, a brain region involved in both seizure activity and memory formation. Investigators are targeting the perforant pathway from EC to hippocampus, which primarily relies of layers II and III of EC. Therefore, this targeting will ensure that layers II and III of EC are within the beam profile of LIFU. During study visits, participant will receive non-invasive ultrasound stimulation in their brains. Investigators will measure seizure frequency and epileptic activity using the implanted RNS system to assess LIFU's effects for epilepsy. Neuropsychological and memory tests will be conducted before and after LIFU application to detect changes in cognitive functions. Investigators will compare results before and after stimulation to determine LIFU's effectiveness in reducing seizures and potentially improving memory or other cognitive functions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of medically refractory focal epilepsy of mesial temporal onset
* RNS system implantation in the hippocampus
* Prior MRI and CT of the head
* Able to consent for themselves
* Internet access

Exclusion Criteria:

* TBI (ongoing, or in the prior 6 months)
* Currently pregnant or breastfeeding
* Progressive diseases - such as autoimmune epilepsies or diagnosis of a progressive neurological disorder
* Status epilepticus within one year of study start
* History of suicidal ideation or attempts in the last 6 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Seizure Frequency | 6 months past their final research study visit
  Utilizing the implanted RNS system patient seizure frequency will be monitored over time following both real and sham intervention.

SECONDARY OUTCOMES:
Report of Symptoms Questionnaires | Within session, approximately over a 3 hour period.
  To evaluate the safety profile and tolerability of LIFU delivery, measured by a series questionnaires pre and post LIFU application evaluating symptoms and side-effects. Participants are asked to report any existing (pre) & new (post) symptoms
Memory Encoding | Within session, over approximately 3 hours.
  To evaluate the cognitive effects of LIFU delivery on memory, participants will be assessed for correct vs incorrect encoding (face/name pair shown, & then queried after a distractor task). % correct will be assessed.
Working Memory Task | Within session, over approximately 3 hours.
  To evaluate the cognitive effects of LIFU delivery on working memory, participants will be assessed for correct vs incorrect encoding (given a list of objects, asked to recall in smallest to largest order). % correct will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Aashit Shah, MD, Principal Investigator — Carilion Clinic
Locations (1):
- Fralin Biomedical Research Institute at VTC, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No